CLINICAL TRIAL: NCT00165490
Title: Phase II Trial of Cetuximab, Irinotecan, Cisplatin (CPC), Concurrent Radiation Therapy, and Surgery for Resectable Esophageal Cancer
Brief Title: Combination Chemotherapy, Radiation Therapy and Surgery for Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Peter C. Enzinger, MD, Overall PI, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-012
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Adenocarcinoma of Esophagus; Squamous Cell Carcinoma of Esophagus
Keywords: adenocarcinoma of esophagus; squamous cell carcinoma of esophagus; combination chemotherapy; cisplatin; irinotecan; radiation therapy; resectable esophageal cancer
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Cetuximab; Cisplatin; Irinotecan; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cetuximab — Given once per week on weeks 1-8 and restarted 4 weeks after surgery, once weekly for 6 months.
Drug: Cisplatin — Given once per week on weeks 1, 2, 4,and 5.
Drug: Irinotecan — Given once per week on weeks 1, 2, 4,and 5.
Device: Radiation therapy — Once daily for 28 treatments (5 1/2 weeks)
Procedure: Surgery — Surgery performed 4-8 weeks after chemoradiation therapy.

SUMMARY:
The purpose of this study is to find out what effects (good and bad) the combination of three chemotherapy drugs (cetuximab, cisplatin, and irinotecan) have on esophageal cancer when given with radiation therapy.

DETAILED DESCRIPTION:
* Patients participating in this study must have a tumor biopsy taken to confirm the type of tumor.
* Outpatient therapy with cetuximab alone will be given intravenously on week 0.
* During week 1-8 outpatient radiation therapy will be started and continued once per day for 28 treatments or 5 1/2 weeks.
* Outpatient chemotherapy (cisplatin, irinotecan and cetuximab) is given once per week on weeks 1, 2, 4, and 5. Cetuximab alone will be given on weeks 3, 6, 7, and 8.
* A repeat CT scan and PET scan will be performed to restage the tumor on week 8. This is to confirm that the cancer has remained localized.
* Inpatient surgery is scheduled 4 to 8 weeks after completion of chemotherapy and radiation therapy.
* Cetuximab will be restarted within 4 weeks after surgery and continue weekly for 6 months.
* During chemotherapy and radiation therapy, physical exams and vital signs will be performed before each chemotherapy treatment. Routine blood tests will also be performed.
* Between chemotherapy-radiation therapy and surgery a CAT scan of chest, abdomen and pelvis along with a PET scan will be performed.
* After surgery a CAT scan of chest, abdomen and pelvis will be performed every 3 months for 2 years then every 6 months for 3 years. An EGD (upper endoscopy) with biopsy will be done every 6 months for 2 years and then yearly for 3 years. Physical exam, vital signs and routine blood tests will be done every 2 weeks for 6 months, then every 3 months for 1.5 years, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Negative pregnancy test
* Adenocarcinoma or squamous cell carcinoma of the esophagus, including the gastroesophageal junction, histologically confirmed, stage IIA, IIB and III.
* ECOG performance status of 0 or 1.
* Neutrophils greater or equal to 1,500/ul
* Platelets greater or equal to 100,000/ul
* Serum bilirubin less or equal to 1.5mg/ul
* Serum creatinine less or equal to 1.5mg/ul
* AST or SGOT less or equal to 2.5x upper normal limit
* Alkaline phosphatase less or equal to 5x upper normal limit

Exclusion Criteria:

* Prior surgery for esophageal or gastro-esophageal junction cancer.
* Prior chemotherapy or radiation therapy
* Biopsy proven tumor invasion of the tracheobronchial tree or tracheo-esophageal fistula.
* Metastatic disease to distant organs or non-regional lymph nodes.
* Co-morbid disease that in the opinion of the investigator makes combined chemo-radiotherapy inadvisable.
* Pregnant or lactating women
* Other active malignancy
* Patients with known Gilbert's Disease or interstitial pulmonary fibrosis.
* History of seizure disorder
* Uncontrolled diarrhea
* Peripheral neuropathy (Grade 2)
* Prior cetuximab or other therapy that specifically and directly targets the EGF pathway.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-08; Primary Completion 2007-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
To determine the response to the combination of cetuximab, cisplatin, irinotecan, and radiation therapy in resectable esophageal carcinoma. | 3 years

SECONDARY OUTCOMES:
To determine the safety of the drug combination and radiation therapy | 3 years
To determine the progression-free survival of patients treated with combination chemotherapy and radiation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Enzinger, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts